CLINICAL TRIAL: NCT06525220
Title: A Phase 3 Randomized, Open-label Study to Evaluate the Efficacy and Safety of Petosemtamab Plus Pembrolizumab vs Pembrolizumab in First-line Treatment of Recurrent or Metastatic PD-L1+ Head and Neck Squamous Cell Carcinoma
Brief Title: A Phase 3 Study to Evaluate Petosemtamab Plus Pembrolizumab vs Pembrolizumab in First-line Treatment of Head and Neck Cancer (LiGeR - HN1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-158-CL03; 2023-510323-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; PD-L1+; Head and Neck cancer; Petosemtamab; Pembrolizumab; Liger; Oral Cavity; Oropharynx; Larynx; Hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Laryngeal Diseases | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Petosemtamab + Pembrolizumab (Experimental): Combination Therapy
  Interventions: Drug: Petosemtamab; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): Monotherapy
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Petosemtamab — MCLA-158
  Arms: Petosemtamab + Pembrolizumab
Drug: Pembrolizumab — Humanized Antibody

SUMMARY:
This is a Phase 3 randomized, open-label study to evaluate the efficacy and safety of petosemtamab plus pembrolizumab vs pembrolizumab in first-line treatment of recurrent or metastatic PD-L1+ head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, open-label study to evaluate the efficacy and safety of petosemtamab plus pembrolizumab vs pembrolizumab in first-line treatment of recurrent or metastatic PD-L1+ HNSCC. HNSCC patients should not have had previous systemic therapy administered in the incurable recurrent or metastatic setting, although previous systemic therapy as part of multimodal treatment for locally advanced disease is allowed if PD was ≥6 months after the last platinum-containing therapy dose. Previous treatments with anti PD-(L)1 or anti-EGFR therapies are not allowed. In the case of cetuximab, patients who have received cetuximab with radiotherapy as a local treatment and PD was >1 year after the last dose of cetuximab are eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF before initiation of any study procedures
2. Age ≥ 18 years at signing of ICF
3. Histologically confirmed HNSCC with evidence of metastatic or locally recurrent disease not amenable to local therapy with curative intent.
4. The eligible HNSCC primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
5. HNSCC patients eligible to receive pembrolizumab as 1L monotherapy with tumors expressing PD-L1, CPS ≥1.
6. HNSCC patients should not have had previous systemic therapy administered in the incurable recurrent or metastatic setting
7. A new tumor biopsy, unless the patient has an available archival tumor sample with sufficient material
8. Measurable disease per Investigator assessment as defined by RECIST v1.1 by radiologic methods
9. ECOG Performance Status (PS) of 0-1
10. Life expectancy ≥ 12 weeks, as per investigator assessment.
11. Left ventricular ejection fraction (LVEF) ≥50% or ≥ institutional normal limit, whichever is higher, by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
12. Adequate organ function as defined per protocol.
13. HIV-positive patients are eligible only if the cluster of differentiation 4 (CD4+) count is ≥ 300/µl, viral load is undetectable, and the patient is currently receiving highly active antiretroviral therapy

Exclusion Criteria:

1. Central nervous system metastases that are untreated or already treated but symptomatic, or require radiation, surgery, or continued steroid therapy to control symptoms within 21 days prior to randomization
2. Known leptomeningeal involvement
3. Any systemic anticancer therapy or investigational drug within 4 weeks or 5 half-lives, whichever is shorter, before randomization
4. Requirement for immunosuppressive medication
5. Major surgery or radiotherapy within 3 weeks of randomization
6. Clinically significant toxicities related to prior anticancer therapies that have not returned to ≤ Grade 1 or baseline except for Grade ≤2- myalgia, neuropathy, alopecia, and any prior therapy related endocrinopathies
7. History of hypersensitivity reaction to any of the excipients of petosemtomab or pembrolizumab.
8. Unstable angina; history of congestive heart failure of Class II-IV New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment; or history of myocardial infarction within 6 months prior to randomization
9. History of prior malignancies within the last 5 years, with the exception of excised local cancer
10. Current dyspnea at rest of any origin, or other diseases requiring continuous oxygen therapy
11. Current serious illness or medical conditions including, but not limited to, uncontrolled active infection, clinically significant pulmonary, metabolic or psychiatric disorders
12. Patients with known infectious diseases as per protocol.
13. Pregnant or breastfeeding patients.
14. The patient has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy of prednisone >10 mg/day or equivalent, or any other form of immunosuppressive therapy
15. The patient has an active autoimmune disease that has required systemic immune suppressive treatment in the past 2 years; replacement therapy is not considered immune suppressive treatment
16. The patient has had an allogeneic tissue/solid organ transplant.
17. Patient has a primary tumor site of nasopharynx, or sinonasal carcinoma (any histology)

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3 years
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by blinded independent central review (BICR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Progression Free Survival (PFS) per RECIST v1.1 as assessed by BICR | Up to approximately 2 years
Duration of Response (DOR) per RECIST v1.1 as assessed by BICR | Up to approximately 2 years
Objective response rate per RECIST v1.1 as assessed by investigator review | Up to approximately 2 years
Progression-free survival per RECIST v1.1 as assessed by investigator review | Up to approximately 2 years
Duration of response per RECIST v1.1 as assessed by investigator review | Up to approximately 2 years
Clinical benefit rate per RECIST v1.1 as assessed by BICR | Up to approximately 2 years
Clinical benefit rate per RECIST v1.1 as assessed by investigator review | Up to approximately 2 years
Number of participants who experienced at least one treatment emergent adverse event (TEAE) | Up to 30 days post last dose
Number of participants who experienced at least one serious TEAE | Up to 30 days post last dose
Number of participants who discontinued study treatment due to TEAEs | Up to 30 days post last dose
Number of participants who had dose modification due to TEAEs | Up to 30 days post last dose
To evaluate patient reported outcomes for health-related quality of life | Up to approximately 2 years
Pharmacokinetic parameters | Up to first 6 cycles
Incidence of anti-drug antibodies (ADAs) | Up to 30 days post last dose

CONTACTS AND LOCATIONS:
Locations (179):
- United States (35):
  - Site 164, Mobile, Alabama
  - Site 36, La Jolla, California
  - Site 27, Los Angeles, California
  - Site 16, Palo Alto, California
  - Site 19, Newark, Delaware
  - Site 108, Washington D.C., District of Columbia
  - Site 14, Fort Myers, Florida
  - Site 48, Orlando, Florida
  - Site 8, Orlando, Florida
  - Site 21, St. Petersburg, Florida
  - Site 20, West Palm Beach, Florida
  - Site 171, Atlanta, Georgia
  - Site 50, Chicago, Illinois
  - Site 2, Louisville, Kentucky
  - Site 162, Baton Rouge, Louisiana
  - Site 155, Minneapolis, Minnesota
  - Site 168, St Louis, Missouri
  - Site 94, Hackensack, New Jersey
  - Site 6, Albuquerque, New Mexico
  - Site 113, Durham, North Carolina
  - Site 118, Winston-Salem, North Carolina
  - Site 43, Philadelphia, Pennsylvania
  - Site 153, Philadelphia, Pennsylvania
  - Site 154, Philadelphia, Pennsylvania
  - Site 89, Chattanooga, Tennessee
  - Site 115, Memphis, Tennessee
  - Site 88, Nashville, Tennessee
  - Site 22, Austin, Texas
  - Site 1, Houston, Texas
  - Site 18, Plano, Texas
  - Site 17, Sugarland, Texas
  - Site 15, Tyler, Texas
  - Site 10, Salt Lake City, Utah
  - Site 12, Blacksburg, Virginia
  - Site 23, Norfolk, Virginia
- Argentina (7):
  - Site 170, CABA
  - Site 96, CABA
  - Site 37, CABA
  - Site 31, Córdoba
  - Site 30, La Rioja
  - Site 76, Rosario
  - Site 46, Viedma
- Australia (4):
  - Site 11, Blacktown, New South Wales
  - Site 24, St Leonards, New South Wales
  - Site 166, Greenslopes, Queensland
  - Site 151, Melbourne, Victoria
- Belgium (6):
  - Site 53, Brussels
  - Site 98, Edegem
  - Site 99, Ghent
  - Site 71, Leuven
  - Site 109, Liège
  - Site 63, Namur
- Brazil (9):
  - Site 149, Rio de Janeiro, Rio de Janeiro
  - Site 141, Belo Horizonte
  - Site 144, Natal
  - Site 140, Porto Alegre
  - Site 142, Porto Alegre
  - Site 137, Recife
  - Site 138, Rio de Janeiro
  - Site 134, São Paulo
  - Site 136, São Paulo
- Canada (3):
  - Site 165, St. John's
  - Site 44, Toronto
  - Site 111, Winnipeg
- Chile (7):
  - Site 38, Antofagasta
  - Site 26, Providencia
  - Site 29, Recoleta
  - Site 40, Santiago
  - Site 32, Santiago
  - Site 34, Santiago
  - Site 25, Temuco
- France (14):
  - Site 56, Bordeaux
  - Site 101, Le Mans
  - Site 79, Lille
  - Site 72, Lyon
  - Site 57, Marseille
  - Site 55, Montpellier
  - Site 66, Nice
  - Site 105, Paris
  - Site 143, Paris
  - Site 87, Poitiers
  - Site 54, Rouen
  - Site 59, Toulouse
  - Site 64, Vandœuvre-lès-Nancy
  - Site 112, Villejuif
- Germany (13):
  - Site 133, Bonn
  - Site 178, Dortmund
  - Site 100, Dresden
  - Site 60, Greifswald
  - Site 82, Hamburg
  - Site 91, Hamburg
  - Site 104, Hanover
  - Site 129, Mannheim
  - Site 148, München
  - Site 121, Münster
  - Site 78, Tübingen
  - Site 130, Ulm
  - Site 110, Würzburg
- Greece (5):
  - Site 119, Pátrai, Achaia
  - Site 156, Athens, Attica
  - Site 117, Heraklion, Crete
  - Site 95, Chaïdári
  - Site 92, Panórama
- Israel (4):
  - Site 9, Haifa
  - Site 5, Jerusalem
  - Site 3, Ramat Gan
  - Site 7, Tel Aviv
- Italy (8):
  - Site 86, Ancona
  - Site 97, Brescia
  - Site 139, Meldola
  - Site 122, Milan
  - Site 81, Milan
  - Site 152, Naples
  - Site 93, Naples
  - Site 85, Rozzano
- Japan (7):
  - Site 167, Nagoya, Aichi-ken
  - Site 123, Kashiwa, Chiba
  - Site 127, Hiragi, Kagawa-ken
  - Site 174, Natori-shi, Miyagi
  - Site 126, Sendai, Miyagi
  - Site 125, Ōsaka-sayama, Osaka
  - Site 124, Chuo Ku, Tokyo
- Site 179, Vilnius, Lithuania
- Malaysia (3):
  - Site 163, Johor Bahru
  - Site 159, Kuching
  - Site 161, Putrajaya
- Netherlands (3):
  - Site 84, Amsterdam
  - Site 58, Nijmegen
  - Site 68, Utrecht
- Poland (5):
  - Site 150, Bydgoszcz
  - Site 131, Gdansk
  - Site 106, Gliwice
  - Site 116, Krakow
  - Site 158, Warsaw
- Portugal (2):
  - Site 172, Coimbra
  - Site 175, Porto
- South Korea (9):
  - Site 145, Busan
  - Site 13, Goyang-si
  - Site 47, Gyeonggi-do
  - Site 51, Hwasun
  - Site 28, Seoul
  - Site 35, Seoul
  - Site 45, Seoul
  - Site 42, Suwon
  - Site 157, Suwon
- Spain (10):
  - Site 120, Badalona
  - Site 80, Barcelona
  - Site 128, Madrid
  - Site 75, Madrid
  - Site 67, Madrid
  - Site 160, Madrid
  - Site 73, Marbella
  - Site 61, Pamplona
  - Site 62, Pamplona
  - Site 74, Valencia
- Taiwan (7):
  - Site 41, Changhua
  - Site 4, Kaohsiung City
  - Site 103, Kaohsiung City
  - Site 52, Taichung
  - Site 39, Taipei
  - Site 33, Taipei
  - Site 49, Taoyuan
- Thailand (5):
  - Site 114, Bangkok Noi, Bangkok
  - Site 107, Pathum Wan, Bangkok
  - Site 65, Ratchathewi, Bangkok
  - Site 146, Chiang Rai, Changwat Chiang Rai
  - Site 77, Hat Yai, Changwat Songkhla
- Site 176, Antalya, Turkey (Türkiye)
- United Kingdom (11):
  - Site 102, Cambridge
  - Site 169, Cardiff
  - Site 132, London
  - Site 90, London
  - Site 69, London
  - Site 173, Manchester
  - Site 177, Newcastle upon Tyne
  - Site 83, Northwood
  - Site 147, Southampton
  - Site 70, Sutton
  - Site 135, Taunton

REFERENCES:
- [Derived] Machiels JP, Fayette J, Haddad R, Adkins D, Gillison M, Harrington KJ, Kim SB, Le Tourneau C, Psyrri A, Rosenberg A, Siu LL, Tahara M, William WN Jr, Ford J, Jauhari S, Pyle R, Shen YM, Yao D, Zohren F, Vokes E. LiGeR-HN phase III trials of petosemtamab + pembrolizumab and petosemtamab monotherapy in recurrent or metastatic HNSCC. Future Oncol. 2025 Jul;21(16):2007-2016. doi: 10.1080/14796694.2025.2511470. Epub 2025 Jun 13. PMID 40511820